CLINICAL TRIAL: NCT04002856
Title: Aesthetic Performance and Tolerance Evaluation of "Profhilo®" Injective Intradermal Treatment for the Skin Roughness and Laxity of the Neck
Brief Title: Aesthetic Performance of "Profhilo®" Injective Intradermal Treatment for the Neck
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Derming SRL (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E0319
Record Dates: First submitted 2019-06-27; First posted 2019-07-01 (Actual); Last update posted 2019-07-18 (Actual); Status verified 2019-06

CONDITIONS: Skin Manifestations
MeSH Terms: conditions — Skin Manifestations

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Profhilo® (Experimental): The 1st treatment was performed during T0 visit, after the basal evaluations planned by the study procedure and repeated after 1 month (T1).
  2 mL of Profhilo® was injected into the middle-deep dermis by needle (29 G) using a bolus technique called "BAP" (Bio Aesthetic Point technique); this technique involves a series of 10 micro-wheals on 3 vertical-lines (3-4-3 ). The amount of product injected was 0.2 ml for each injection point.
  Interventions: Device: Profhilo®

INTERVENTIONS:
Device: Profhilo® — Profhilo® (IBSA Farmaceutici Italia S.r.l.) is a resorbable medical device 2.25 ml non-pyrogenic pre-filled syringe, containing 2 ml of 3.2% hyaluronic acid for intradermal use (32 mg H-HA + 32 mg L-HA dissolved in 2 ml of saline buffered sodium chloride

SUMMARY:
The objective of this study is to investigate the aesthetic performance of the Hyaluronic acid (HA)-based dermal filler Profhilo® injected by a novel bio aesthetic point technique ("BAP" techinique ) in woman aged 40-65 years with skin flaccidity and roughness of the neck.

ELIGIBILITY:
Inclusion Criteria:

* female sex,
* 40-65 years,
* 3-4 neck roughness/laxity grade according to a clinical reference scale;
* asking for neck laxity and roughness restoration;
* available and able to return to the study site for the post-procedural follow-up examinations;
* accepting to not change their habits regarding food, physical activity, cosmetic and cleansing products for the neck;
* accepting to not expose their neck to strong UV irradiation (UV session, or sun bathes) during the entire duration of the study, without appropriate sun protection;
* accepting to sign the informed consent form.

Exclusion Criteria:

* Pregnancy;
* lactation;
* smokers;
* alcohol abuse and/or drug use;
* subjects not in menopause who do not use adequate contraceptive precautions in order to avoid pregnancies during the study;
* subjects not in menopause who do not accept to perform the pregnancy test at T0 (before the 1st aesthetic procedure) and at T1 (1 month after the 1st injection treatment execution, before the 2nd aesthetic procedure);
* Body Mass Index (BMI) variation (± 1) during the study period;
* performing skin treatments for neck aesthetic correction (biomaterials implants, neck lifting, botox injections, laser, chemical peeling) in the 6 months prior to the study start;
* performing permanent filler in the past;
* change in the normal habits regarding food, physical activity, neck cosmetic and cleansing use during the month preceding the test;
* sensitivity to the test product or its ingredients (to be assessed by the investigator during the baseline visit);
* subjects whose insufficient adhesion to the study protocol is foreseeable;
* participation in a similar study currently or during the previous 9 months;
* dermatitis;
* presence of cutaneous disease on the tested area, as lesions, scars, malformations;
* recurrent facial/labial herpes;
* clinical and significant skin condition on the test area (e.g. active eczema, psoriasis, severe rosacea, scleroderma, local infections and severe acne);
* diabetes;
* endocrine disease;
* hepatic disorder;
* renal disorder;
* cardiac disorder;
* pulmonary disease;
* cancer;
* neurological or psychological disease;
* inflammatory/immunosuppressive disease;
* drug allergy;
* Anticoagulants and antiplatelet drugs, anti-histaminic, topic and systemic corticosteroids, narcotic, antidepressant, immunosuppressive drugs (with the except of contraceptive or hormonal treatment starting more than 1 year ago);
* using of drugs able to influence the test results in the investigator opinion.

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2019-02-18 (Actual); Primary Completion 2019-06-21 (Actual); Study Completion 2019-06-21 (Actual)

PRIMARY OUTCOMES:
Change from baseline of neck skin roughness and laxity clinical grade | Baseline (T0), 1 month (T1), 4 months (T2)
  Skin roughness and laxity clinical grade, according to a visual score from 1 (no roughness and flaccidity) to 5 (very severe roughness and flaccidity).
Change from baseline of superficial skin hydration | Baseline (T0), 1 month (T1), 4 months (T2)
  Skin electrical capacitance value was measured mono-laterally on the neck with Corneometer CM825 (Courage - Khazaka, Köln, Germany). The measure of the skin capacitance properties is an indirect expression of its hydration level.
Change from baseline of deep skin hydration | Baseline (T0), 1 month (T1), 4 months (T2)
  Tissue dielectric constant value of superficial and deep skin layers was measured mono-laterally on the neck with MoistureMeterD (Delfin Technologies, Kuopio - Finland)
Change from baseline of skin density | Baseline (T0), 1 month (T1), 4 months (T2)
  A little skin area of about 7 cm2 at level of neck was pinched, in standardized conditions, using a specific device. Because of this "pinch" the skin profile changes depending on cutaneous density; when the skin is slack the "pinch" forms a lot of wrinkles. A picture of the skin pinched was taken thanks to Primos compact portable device (GFMesstechnik); Primos software is able to measure skin principal profilometric parameters.
Change from baseline of skin plastoelasticity | Baseline (T0), 1 month (T1), 4 months (T2)
  Superficial and deep skin plastoelasticity was measured mono-laterally on the neck with the instrument Dermal Torque Meter (Dia-Stron Ltd., UK).
Change from baseline of photographic documentation | Baseline (T0), 1 month (T1), 4 months (T2)
  2D pictures of the neck

CONTACTS AND LOCATIONS:
Locations (1):
- DERMING, Milan, MI, Italy